CLINICAL TRIAL: NCT02886754
Title: The Effect of a Proficiency Based Progression Training Programme for Clinical Communication on ISBAR Performance
Brief Title: Proficiency-Based Progression Training for Clinical Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dorothy Breen, Specilaist in Intensive Care and Director of Education, ASSERT, Principal Invesitgator, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ISBAR
Record Dates: First submitted 2016-08-27; First posted 2016-09-01 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Clinical Communication; ISBAR; Simulation; Proficiency-Based Progression; Non Technical Skills; Performance; Deteriorating Patient
Keywords: Clinical Communication; ISBAR; Simulation; Performance; Non technical skills; Proficiency

STUDY DESIGN:
Intervention Model Description: The study design is a parallel group, double-blind, randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors were unaware of which intervention group subjects were allocated
Oversight: Data Monitoring Committee: No

ARMS (3):
- National e-learning programme only (HSE) (Active Comparator): National e-learning programme only Recent successful completion the National e-learning programme by certificate will be displayed. Students then complete a student satisfaction survey and proceed directly for performance assessment to the high-fidelity simulation suite.
  Interventions: Behavioral: National e-learning programme only
- Simulation (S) (Active Comparator): Simulation Recent successful completion of the National e-learning e-learning programme by certificate will be displayed. Students will proceed to standard simulation using the same series of paper cases as PBP which prompt simulated phone calls but no requirement to meet a proficiency benchmark. 4 hours will be allotted to this training. Following training participants will complete the student satisfaction survey and will then proceed directly for performance assessment to the high-fidelity simulation suite.
  Interventions: Behavioral: National e-learning programme only; Behavioral: Standard simulation
- Proficiency-Based Progression (PBP) (Experimental): Recent successful completion of the National e-learning programme by certificate will be displayed. Students will proceed to PBP simulation using the same series of paper cases as S which prompt simulated phone calls. PBP students will be scored according to predefined metrics and will be required to reach proficiency benchmarks. Following training participants will complete the student satisfaction survey and proceed directly for performance assessment to the high-fidelity simulation suite.
  Interventions: Behavioral: Proficiency-based progression; Behavioral: National e-learning programme only

INTERVENTIONS:
Behavioral: Proficiency-based progression — Use of validated metrics and performance benchmarks to simulation training
  Other Names: PBP
  Arms: Proficiency-Based Progression (PBP)
Behavioral: National e-learning programme only — National e-learning programme (COMPASS)
  Other Names: HSE
Behavioral: Standard simulation — Paper based simulation cases
  Other Names: Simulation S
  Arms: Simulation (S)

SUMMARY:
Importance: Clinical communication is an important source of medical error and preventable adverse events.

Objective: To determine the effectiveness of proficiency-based progression (PBP) simulation training for ISBAR (Identify, Situation, Background, Assessment, Recommendation) communication in the deteriorating patient.

Setting: The study will be conducted in University College Cork, Ireland. Participants: Third year undergraduate nursing and fifth year medical students, who are scheduled to undertake ISBAR training as part of the National Early Warning Score (NEWS) programme.

Intervention: Participants will be prospectively randomized to one of three groups before undertaking a performance assessment of an ISBAR communication relevant to a deteriorating patient in a high fidelity simulation laboratory: HSE group (the national e-learning programme only); S group (national e- learning plus simulation training) and PBP group (national e-learning plus proficiency-based progression simulation).

Main outcome and measures: A proficiency benchmark on the performance of ISBAR communication in the context of an acutely deteriorating patient.

DETAILED DESCRIPTION:
The first successful simulation validation study used a proficiency-based progression methodology. Since then the approach has been successfully deployed to produce superior technical skills but has not yet been validated for non-technical (communication) skills. The ISBAR (Identify, Situation, Background, Assessment and Recommendation) has been selected as the standardised tool for clinical communication in relation to an acutely deteriorating patient in many healthcare organisations worldwide, including Ireland.

The aim of this study is to explore whether proficiency-based progression (PBP) could be applied to simulation-based training for ISBAR performance to produce a superior skill set.

The study will compare performance outcomes of students, who receive the national e-learning programme only with those who receive it in combination with either standard simulation or proficiency-based progression (PBP) simulation.

Participants will be prospectively randomized to one of three training groups within their professional cohort (medicine or nursing) before undertaking a performance assessment of an ISBAR communication relevant to a deteriorating patient in a high fidelity simulation laboratory:

1. Online learning only (HSE) -the national e-learning programme only
2. Standard simulation (S) -online learning plus simulation training
3. Proficiency based progression (PBP) -online learning plus proficiency-based progression simulation.

Main outcome and measures: A proficiency benchmark on the performance of ISBAR communication in the context of an acutely deteriorating patient.

All participants will be required to demonstrate a certificate of successful completion on the national e-learning programme within the previous 4 weeks as well as supplying baseline demographic information before undertaking the training.

Performance metrics have previously been identified, operationally defined and agreed upon at a modified Delphi panel meeting consisting of medical and nursing experts for a series of paper-based simulation cases and a standardised high fidelity simulation case used as the assessment case. The proficiency benchmark for each case has been set based on the performance of experienced nursing and medical personnel on each case as a series of steps, errors and critical errors.

Outcome assessment will be scored by reviewing recordings of ISBAR performance by each participant on the standardised case in the high fidelity laboratory.

ELIGIBILITY:
Inclusion Criteria:

Third year undergraduate nursing students

Fifth year medical students

Exclusion Criteria:

Lack of consent

Failure to successfully complete the National e-learning NEWS programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
Proportion of those reaching the benchmark on the assessment case | 6 months
  Independent review by two blinded assessors of recorded ISBAR phone call conducted in the high fidelity simulation setting

SECONDARY OUTCOMES:
Number of completed steps | 6 months
  Number of successfully completed steps as predefined by the metrics for the assessment case

OTHER OUTCOMES:
Number of total errors | 6 months
  Number of total errors as predefined by the metrics for the assessment case
Number of errors/critical errors | 6 months
  Number of errors/critical errors as predefined by the metrics for the assessment case

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gallagher, PhD, DSc, Study Director — University College Cork, College Rd, Cork Ireland
Locations (1):
- University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gallagher AG, Seymour NE, Jordan-Black JA, Bunting BP, McGlade K, Satava RM. Prospective, randomized assessment of transfer of training (ToT) and transfer effectiveness ratio (TER) of virtual reality simulation training for laparoscopic skill acquisition. Ann Surg. 2013 Jun;257(6):1025-31. doi: 10.1097/SLA.0b013e318284f658. PMID 23426342
- [Background] Angelo RL, Ryu RK, Pedowitz RA, Beach W, Burns J, Dodds J, Field L, Getelman M, Hobgood R, McIntyre L, Gallagher AG. A Proficiency-Based Progression Training Curriculum Coupled With a Model Simulator Results in the Acquisition of a Superior Arthroscopic Bankart Skill Set. Arthroscopy. 2015 Oct;31(10):1854-71. doi: 10.1016/j.arthro.2015.07.001. Epub 2015 Sep 2. PMID 26341047
- [Background] Van Sickle KR, Ritter EM, Baghai M, Goldenberg AE, Huang IP, Gallagher AG, Smith CD. Prospective, randomized, double-blind trial of curriculum-based training for intracorporeal suturing and knot tying. J Am Coll Surg. 2008 Oct;207(4):560-8. doi: 10.1016/j.jamcollsurg.2008.05.007. Epub 2008 Jul 14. PMID 18926460
- [Derived] Breen D, O'Brien S, McCarthy N, Gallagher A, Walshe N. Effect of a proficiency-based progression simulation programme on clinical communication for the deteriorating patient: a randomised controlled trial. BMJ Open. 2019 Jul 9;9(7):e025992. doi: 10.1136/bmjopen-2018-025992. PMID 31289064